CLINICAL TRIAL: NCT07395115
Title: Factors Affecting Optic Nerve Sheath Diameter and Visual Acuity Changes in Adult Patients Undergoing Prone Spine Surgery: A Prospective Observational Study
Brief Title: A Prospective Observational Study on Factors Affecting Optic Nerve Sheath Diameter and Visual Acuity in Prone Spinal Surgery
Acronym: PRONE-ONSD
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Begüm Ramakan, MD, Resident Physician in Anesthesiology and Reanimation, Istanbul University - Cerrahpasa
Other Study IDs: 2024/244
Record Dates: First submitted 2025-12-03; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Spinal Surgery; Prone Position
Keywords: logMAR; Snellen; visual acuity; ONSD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prone Spine Surgery Cohort: Adults undergoing prone-position spine surgery, evaluated with ultrasound ONSD measurements and visual acuity testing.

SUMMARY:
The prone position in spinal surgery can alter intracranial pressure and optic nerve sheath diameter (ONSD) and potentially lead to visual complications. This prospective observational study aimed to identify factors influencing ultrasonographic ONSD changes and visual acuity in patients undergoing spinal surgery.

DETAILED DESCRIPTION:
During spine surgery, many patients are positioned face-down (prone position) for several hours. This position may influence blood flow to the head and increase pressure around the brain and eyes. One structure that can reflect these pressure changes is the optic nerve sheath, which surrounds the optic nerve at the back of the eye. When the pressure inside the skull rises, the optic nerve sheath may become wider. This change can be measured non-invasively using ultrasound and is referred to as optic nerve sheath diameter (ONSD).

This prospective observational study will evaluate whether ONSD changes occur in adult patients undergoing prone-position spine surgery and whether these changes are related to temporary alterations in vision. Visual acuity will be evaluated using a standard Snellen chart before surgery and on the first postoperative day to detect any change in vision after the procedure.

Ultrasound ONSD measurements will be performed in three stages: before the patient is placed in the prone position, shortly after the prone position is established, and at the end of the surgery while still in the same position. Clinical variables such as blood pressure, carbon dioxide levels, ventilation parameters, anesthesia technique, the use of a pinned head holder, and patient characteristics will also be recorded. By comparing these variables with ONSD and visual outcomes, the study aims to identify whether specific surgical or physiological factors contribute to increased optic nerve sheath width or temporary vision disturbances.

This research does not involve any experimental drug or device. All measurements are part of routine safe monitoring techniques used to assess patients' condition during surgery. The goal of this study is to help better understand factors that may increase the risk of eye-related complications during prone spine surgery and to contribute to safer surgical practices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled to undergo elective spine surgery in the prone position
* American Society of Anesthesiologists (ASA) physical status I-III
* Preoperative visual acuity measurable using a Snellen chart

Exclusion Criteria:

* Preexisting ophthalmologic diseases affecting optic nerve or visual acuity (e.g., glaucoma, optic neuropathy, diabetic retinopathy)
* Previous eye trauma or history of orbital surgery
* Inability to obtain reliable ultrasonographic ONSD measurements (e.g., orbital deformity, ocular infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective spine surgery requiring prone positioning at a university hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change in ultrasonographic optic nerve sheath diameter (mm) | Baseline (preoperative, supine), after prone positioning (15 minutes after positioning), and at the end of surgery (intraoperative, before repositioning to supine).
  Optic nerve sheath diameter (ONSD) will be measured bilaterally using standardized transorbital ultrasonography with a high-frequency linear probe (6-13 MHz). Measurements will be obtained 3 mm posterior to the globe, in accordance with established sonographic guidelines. For each eye, three measurements will be recorded, and the mean value will be calculated. The average of both eyes will be used for statistical analysis. The primary outcome will be the absolute change in ONSD (ΔONSD, mm) between baseline and intraoperative prone measurements.

SECONDARY OUTCOMES:
Change in visual acuity (logMAR) | Baseline (preoperative) and postoperative day 1.
  Visual acuity will be initially recorded in decimal format using a standard Snellen chart and subsequently converted to logMAR units for statistical analysis. The outcome will be the absolute change in visual acuity (ΔlogMAR) from baseline to postoperative day 1 (postoperative logMAR minus baseline logMAR).
Correlation between change in ONSD and intraoperative end-tidal carbon dioxide (EtCO₂) | Intraoperative period: baseline (supine), after prone positioning (15 minutes), and at the end of surgery.
  Correlation analysis will be performed between changes in ONSD (ΔONSD, mm) and intraoperative end-tidal carbon dioxide levels (EtCO₂, mmHg) recorded simultaneously with ONSD measurements.
Difference in ONSD change between pinned head holder and non-pinned positioning | ntraoperative period: baseline (supine), after prone positioning (15 minutes), and at the end of surgery.
  Change in ONSD (mm) will be compared between patients positioned using a pinned head holder and those positioned without pin fixation. The outcome will be the between-group difference in ONSD change (mm).
Association between postoperative visual acuity change and intraoperative ONSD change | Baseline (preoperative) and postoperative day 1.
  The association between postoperative change in visual acuity (ΔlogMAR) and intraoperative change in optic nerve sheath diameter (ΔONSD) will be evaluated using regression analysis. Visual acuity will be recorded in decimal format and converted to logMAR for statistical analysis. ONSD will be measured using standardized transorbital ultrasonography and expressed in millimeters.
Correlation between change in ONSD and intraoperative mean arterial pressure (MAP) | Intraoperative period: baseline (supine), after prone positioning (15 minutes), and at the end of surgery.
  Correlation analysis will be performed between changes in ONSD (ΔONSD, mm) and intraoperative mean arterial pressure (MAP, mmHg) recorded simultaneously with ONSD measurements.
Correlation between change in ONSD and intraoperative arterial partial pressure of carbon dioxide (PaCO₂) | Intraoperative period: baseline (supine), after prone positioning (15 minutes), and at the end of surgery.
  Correlation analysis will be performed between changes in ONSD (ΔONSD, mm) and arterial partial pressure of carbon dioxide (PaCO₂, mmHg) obtained from arterial blood gas analysis and recorded simultaneously with ONSD measurements.
Correlation between change in ONSD and intraoperative arterial partial pressure of oxygen (PaO₂) | Time Frame: Intraoperative period: baseline (supine), after prone positioning (15 minutes), and at the end of surgery.
  Correlation analysis will be performed between changes in ONSD (ΔONSD, mm) and arterial partial pressure of oxygen (PaO₂, mmHg) obtained from arterial blood gas analysis and recorded simultaneously with ONSD measurements.
Correlation between change in ONSD and intraoperative positive end-expiratory pressure (PEEP) | Intraoperative period: baseline (supine), after prone positioning (15 minutes), and at the end of surgery.
  Correlation analysis will be performed between changes in ONSD (ΔONSD, mm) and intraoperative positive end-expiratory pressure levels (PEEP, cmH₂O) recorded simultaneously with ONSD measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Korkmaz Dilmen, MD, Prof, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty; Begüm Ramakan, MD, Anesthesiology Resident, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpaşa, Cerrahpaşa Faculty of Medicine Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because individual-level data are not permitted to be disclosed under the current ethical approval.